CLINICAL TRIAL: NCT03437824
Title: Vitamin B12 Treatment in Singers - Assessment of Effects Exploratory Pilot Study
Brief Title: Effects of Vitamin B12 Treatment in Singers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael Johns, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: APP-16-06647
Record Dates: First submitted 2017-07-02; First posted 2018-02-19 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyanocobalamin (Experimental): Vitamin B12, 1,000 mg, Once
  Interventions: Drug: Cyanocobalamin
- Placebo (Placebo Comparator): Normal Saline Solution (0.9% Sodium Chloride), Once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyanocobalamin — 1,000 mg, Once
  Other Names: Vitamin B12
  Arms: Cyanocobalamin
Drug: Placebo — 0.9% Sodium Chloride, Once
  Other Names: Normal Saline Solution
  Arms: Placebo

SUMMARY:
In this study, the investigators aim to assess if vitamin B12 treatment demonstrates a beneficial effect on voice performance. If so, they wish to examine the relationship between the vitamin B12 treatment and the study participant's general well-being.

DETAILED DESCRIPTION:
Through the investigators' experience, they have observed that amongst singers and voice professionals, there is a common belief that there are voice benefits from cobalamin treatment. Consequently, some singers and voice professionals tend to ask for cobalamin injections in order to enhance their vocal performance. However, there are no previous reports that illustrate the effects of vitamin B12 deficiency or treatment on voice performance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years old
* An active singer who is presently singing
* Willing and able to comply with the study requirements
* Completed and signed an informed consent form.

Exclusion Criteria:

* Known vitamin B12 deficiency
* Active or recent vitamin B12 treatment (the subject must not receive vitamin B12 treatment for at least 4 weeks)
* Any known bleeding disorder
* Any known laryngeal pathology
* Plans to start any new treatment, oral/parenteral anticoagulant, supplement, or medication during the study period
* Scored above the highest 10 percentile of performance in all three voice evaluation questionnaires will be withdrawn from the study before the first injection (i.e., scored less than or equal to 7 in the Voice Fatigue Index (VFI), less than or equal to 6 in the Evaluation of the Ability to Sing Easily (EASE), and less than or equal to 4 in the Singing Voice Handicap Index 10 (SVHI-10))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Ability to Sing Easily (EASE) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  1 = Not at All, 2 = Mildly, 3 = Moderately, 4 = Extremely
Singing Voice Handicap Index-10 (SVHI-10) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Almost Always, 4 = Always
0-10 Visual Analog Scale (VAS) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  The scale asks, "How confident are you that your voice will do what you need it to do right now?"; 0 = Not Confident At All, 10 = Extremely Confident
Vocal Fold Swelling (Bastian et al., 2009) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  Happy Birthday, Staccato, Trill; 1 = Poor, 5 = Average, 10 = Excellent
Voice Fatigue Index (VFI) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Almost Always, 4 = Always

SECONDARY OUTCOMES:
Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  1 = Not at All, 5 = Extremely
Patients Health Questionnaire-9 for Depression - Change | Baseline, 1 Hr Post-Injection, 3 Hrs Post-Injection, 24 Hrs Post-Injection, 72 Hrs Post-Injection, 1 Wk Post-Injection
  0 = Not at All, 3 = Extremely

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Shoffel-Havakuk, MD, Study Director — University of Southern California
Locations (1):
- Keck Medicine of USC - Downtown Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Shoffel-Havakuk H, Lava CX, Reuven Y, Moog D, Odell K, Reder LS, Hapner ER, Johns MM 3rd. Effect of Vitamin B12 Injection on the Vocal Performance of Professional Singers: A Randomized, Double-blind, Placebo-Controlled, Crossover Trial. JAMA Otolaryngol Head Neck Surg. 2021 Jan 1;147(1):9-15. doi: 10.1001/jamaoto.2020.4026. PMID 33180098